CLINICAL TRIAL: NCT02183831
Title: Comparison of Clinical Outcomes After Cataract Surgery With and Without Capsular Tension Ring
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 1-2014-0010
Record Dates: First submitted 2014-06-23; First posted 2014-07-08 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-06

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Capsular tension ring non insertion group: The patients who had same cataract surgery procedure without CTR insertion
- Capsular tension ring insertion group: The patients who underwent capsular tension ring insertion just before IOL implantation during cataract surgery
  Interventions: Device: Insertion of the capsular tension ring

INTERVENTIONS:
Device: Insertion of the capsular tension ring
  Other Names: a pre-loaded CTR in single use injector was inserted just before IOL implantation during cataract surgery
  Groups: Capsular tension ring insertion group

SUMMARY:
This study was set up to identify clinical outcomes including a refractive shift or change in IOL calculation accuracy and optical quality after Ophtec® capsular tension ring in the eyes without zonular instability.

ELIGIBILITY:
Inclusion Criteria:

1. age between 40 and 79 years
2. no history of eye surgery or glaucoma
3. a transparent central cornea
4. pupil dilation at the preoperative examination of at least 6.0 mm
5. absence of biomicroscopic signs of pseudoexfoliation
6. normal fundus examination

Exclusion Criteria:

1. presence of ocular disease that might affect the visual outcome (e.g., color vision disturbance, chronic uveitis)
2. presence of ocular disease that might affect contrast sensitivity function (e.g., glaucoma, maculopathy, high myopia)

Ages: 40 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients who were planned to undergo the cataract surgery in Department of Ophthalmology, Yonsei University College of Medicine
Sampling Method: Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2014-05; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Best corrected visual acuity | 1 month after capsular tension ring and intraocular lens implantation (cataract surgery) using capsular tension ring
  Visual acuity measurement using refractive error correction
refractive error | 1 month after capsular tension ring and intraocular lens implantation (cataract surgery) using capsular tension ring
  Autokeratometry (KR-7100; Topcon, Tokyo, Japan) and manifested refraction were performed to examine refractive errors
Anterior chamber depth | 3 months after capsular tension ring and intraocular lens implantation (cataract surgery) using capsular tension ring
  obtained with a Scheimpflug imaging system (Pentacam; OCULUS Optikgeräte GmbH, Wetzlar, Germany)
Ocular aberrations | 1month after capsular tension ring and intraocular lens implantation (cataract surgery) using capsular tension ring
  measured using the ray-tracing aberrometer (iTrace, Tracey Technologies, Houston, TX, USA) at a pupil size of 5 mm in mesopic conditions, without pharmacologic dilatation

SECONDARY OUTCOMES:
constrast sensitivity | 3 months after capsular tension ring and intraocular lens implantation (cataract surgery) using capsular tension ring
  measured at five spatial frequencies (1.5, 3, 6, 12, and 18 Hz) using the Optec 6500 vision testing system
posterior capsular opacity grades | 3 months after capsular tension ring and intraocular lens implantation (cataract surgery) using capsular tension ring
  graded after dilation of pupil over 6 mm, based on slit lamp examination findings
Best corrected visual acuity | 3 months after capsular tension ring and intraocular lens implantation (cataract surgery) using capsular tension ring
  Visual acuity measurement using refractive error correction
refractive error | 3 months after capsular tension ring and intraocular lens implantation (cataract surgery) using capsular tension ring
  Autokeratometry (KR-7100; Topcon, Tokyo, Japan) and manifested refraction were performed to examine refractive errors
Ocular aberrations | 3 months after capsular tension ring and intraocular lens implantation (cataract surgery) using capsular tension ring
  measured using the ray-tracing aberrometer (iTrace, Tracey Technologies, Houston, TX, USA) at a pupil size of 5 mm in mesopic conditions, without pharmacologic dilatation